CLINICAL TRIAL: NCT00446732
Title: Catheter Associated Urinary Tract Infections
Brief Title: The Use of the UroShield Device in Patients With Indwelling Urinary Catheters
Acronym: CAUTI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanovibronix (Industry)
Collaborators: Shaare Zedek Medical Center (Other)
Responsible Party: Dr. Harold Jacob CEO, NanoVibronix
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: US-71-003
Record Dates: First submitted 2007-03-11; First posted 2007-03-13 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Device: UroSshield
- 2 (No Intervention)

INTERVENTIONS:
Device: UroSshield — Attachment of the UroShield device to the external part of the urinary catheter
  Arms: 1

SUMMARY:
According to the Israeli Ministry of Health requirement, this study was designed to evaluate the efficacy of the UroShield system is patients that require urinary catheterization. This was designed to compare standard treatment (urinary catheter alone) with the UroShield treatment in occurrence of catheter associated Urinary Tract infection, pain, discomfort, Biofilm prevention and trauma.

DETAILED DESCRIPTION:
This study is aimed at assessing the effectiveness of the NanoVibronix™ UroShield™ System in comparison to Urinary catheter alone in patients requiring urinary catheterization.

1. Primary objectives

   * To observe the effect of UroShield in reduction of patient's complaints relating to indwelling Urinary Catheters

     * Pain
     * Discomfort
   * To observe the effect of UroShield in the reduction/prevention of Biofilm
   * To observe the effect of UroShield on the occurrence of bacteriuria and/or UTI's on patients with Indwelling Urinary Catheters
2. Safety Objective To assess the safety parameters of the UroShield system
3. Secondary Objectives

   * To observe the effect of UroShield in reduction of Foley Catheter related pain medication in patients with Indwelling Urinary Catheters
   * To observe the effect of UroShield in reduction of antibiotic medication in patients with Indwelling Urinary Catheter
   * To observe the effect of UroShield on the clogging of Urinary Catheter when used chronically and the need to replace the catheter
   * To observe the effect of UroShield on the decrease of Tissue damage of patients with Indwelling Urinary Catheters by measuring cell count before and after removal of catheter

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients age 18 years or older
* Patients requiring or having catheterization for more than 24 hours
* Patient able, agrees and signs the Informed Consent Form

Exclusion Criteria:

* Pregnant or breastfeeding women. Women of child bearing potential will perform a pregnancy test before inclusion into the study
* Presence of any clinically relevant known urinary tract infection
* Patient with condition who is not expected to survive the study period
* Known HIV positive
* Patient has any condition, which precludes compliance with study and/or device instructions.
* Patient is currently participating in another clinical study.
* Known allergy to latex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-04 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
primary end points | up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Shenfeled, MD, Principal Investigator — Sharei Zedek
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel